CLINICAL TRIAL: NCT03708354
Title: Tocotrienols Supplementation for Postmenopausal Women With Low Muscle Strength
Brief Title: Tocotrienols for Skeletal Muscle Health
Acronym: VitE-muscle
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulties in Recruiting
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: L19-011
Record Dates: First submitted 2018-10-10; First posted 2018-10-17 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Dynapenia; Postmenopausal Women
Keywords: skeletal muscle strength
MeSH Terms: interventions — Olive Oil; Tocotrienols

STUDY DESIGN:
Intervention Model Description: dietary supplement
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo softgels will be of the same size/color as the active softgels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): One 430 mg olive oil softgel daily for 24 weeks. Each placebo softgel of 430 mg olive oil will contain no tocotrienol or tocopherols at detectable levels.
  Interventions: Drug: placebo softgel
- Intervention (Active Comparator): One 430 mg tocotrienol softgel daily for 24 weeks. Each tocotrienol softgel (DeltaGold® Tocotrienol 70%) contains 430 mg tocotrienol (90% δ-tocotrienol+10% γ-tocotrienol) with a 70% purity, representing 300 mg tocotrienol.
  Interventions: Drug: DeltaGold® Tocotrienol 70%

INTERVENTIONS:
Drug: placebo softgel — One 430 mg olive oil softgel daily for 24 weeks. Each placebo softgel of 430 mg olive oil will contain no tocotrienol or tocopherols at detectable levels.
  Other Names: olive oil
  Arms: Control
Drug: DeltaGold® Tocotrienol 70% — Each TT softgel (DeltaGold® Tocotrienol 70%) contains 430 mg TT (90% δ-TT+10% γ-TT) with a 70% purity, representing 300 mg TT.
  Other Names: tocotrienol
  Arms: Intervention

SUMMARY:
Sarcopenia, defined as a reduction in muscle mass and strength, is a major health concern for postmenopausal women. Evidence suggests that lowering inflammation levels is an important strategy to help mitigate age-related muscle dysfunction and loss. In this pilot study, the investigators will study a tocotrienol (vitamin-E isomer) intervention for feasibility and quantify its effects on postmenopausal women with low muscle strength. A double blind, placebo controlled trial will be conducted on fifty-two qualified subjects. The participants will be assigned to placebo or tocotrienols for 24 weeks. All participants will receive an Omron Alvita Optimized Pedometer. The investigators will measure muscular endurance, strength, and size and gut microbiome profiles at 0, 12, and 24 weeks. In addition, the investigators will measure serum and muscle inflammatory levels at 0 and 24 weeks. All data will be analyzed statistically at p<0.05.

DETAILED DESCRIPTION:
Sarcopenia is a major health issue in postmenopausal women (PMW). The long-term goal is to develop a new strategy featuring a dietary supplement for alleviating sarcopenia in postmenopausal women. The objective is to test a dietary supplement intervention (delta-tocotrienols, TT) for feasibility, and to quantitatively assess its effects on postmenopausal women with sarcopenia. Due to the limited budget, the investigators will not assess appendicular muscle mass in this pilot study and will focus on muscle strength and function. The central hypotheses are that (i) TT supplementation will alleviate age-associated skeletal muscular dysfunction of postmenopausal women with low muscle strength, and (ii) such changes in skeletal muscle are associated with lowered oxidative stress and inflammation wherein the targets are oxylipins (OxL) and endocannabinoids (eCB), and possible modification of gut microbiota. This is a randomized double-blinded placebo-controlled trial. Fifty-two qualified subjects will be assigned to placebo or TT for 24 weeks. There are 4 specific aims (SA) in this study. SA 1 is to evaluate the effects of TT intervention on endurance, strength, function and size of the lower-extremity musculature in PMW with low muscle strength. SA 2 is to measure the effects of TT intervention on oxidative stress and inflammatory levels. SA 3 is to measure the effects of TT intervention on inflammatory OxL and eCB levels in plasma and muscle tissue. SA 4 is to evaluate the effects of TT intervention on abundance and composition of intestinal bacterial in feces. The outcome measures of SA 1 will be assessed at the baseline, after 12 and 24 weeks. The outcome measures of SA 2, SA 3, and SA 4 will be assessed at the baseline and after 24 weeks. In addition, at 0 and 24 weeks, the investigators will monitor (i) compliance by pill count and (ii) changes in lifestyle throughout the study via food intake surveys and physical activity surveys. Descriptive statistics, bivariate tests, and general/generalized linear mixed modeling will be used for the quantitative analysis on the effects of the TT intervention.

ELIGIBILITY:
Inclusion criteria:

1. Postmenopausal women (60-85 yr) not on hormone replacement therapy in the past year.
2. Normal liver, kidney, thyroid function (TSH), serum 25-OH vitamin D (≥ 20 ng/ml)-sent to Quest Diagnostic Laboratory.
3. Grip strength weakness (<20 kg).
4. Sedentary -evaluated by using self-administered International Physical Activity Questionnaire (IPAQ) short form.

Exclusion criteria:

1. Serious chronic disease (e.g., unstable CVD, uncontrolled diabetes, uncontrolled hypertension, active cancer, Parkinson's disease).
2. Taking hormone replacement therapy within 3 months before study starts.
3. Taking medications (i.e., steroids) within 3 months before study starts, since steroids could affect muscle function.
4. Taking supplements (i.e., fish oil) that have anti-inflammatory action during the past 3 months.
5. Having dementia or other medical/eating disorder (i.e. currently receiving an appetite stimulant).
6. Self-report of >10% body weight loss in the past month.
7. Taking anticoagulants that may interact with tocotrienols.

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Aging and decline of estrogen are factors that contribute to skeletal muscle disorders in postmenopausal women.
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
lower-body muscle endurance | 24 weeks
  assessed by 6-min walk test

SECONDARY OUTCOMES:
8-OHdG | 24 weeks
  urine 8-hydroxy-2'-deoxyguanosine
oxylipins | 24 weeks
  oxylipins levels in plamsa and skeletal muscle biopsy
gut microbiome | 24 weeks
  abundance and composition of intestine microbiome in feces
handgrip strength | 24 weels
  assessed by a hand dynamometer
lower-body muscle strength | 24 weeks
  assessed by isometric knee extension muscle strength
functional performance | 24 weeks
  assessed by Time Up and Go test
Muscle size of the lower-extremity musculature | 24 weeks
  cross-sectional area of the rectus femoris assessed using a diagnostic ultrasound device
F2-isoprostanes | 24 weeks
  F2-isoprostanes in urine
TNF-alpha | 24 weeks
  Transforming necrosis factor-alpha in urine
hs-CRP | 24 weeks
  high sensitivity C-reactive protein
endocannabinoid | 24 weeks
  endocannabinoid levels in plasma and muscle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Chwan-Li Shen, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No